CLINICAL TRIAL: NCT04940858
Title: Evaluation of Dentists Burnout in Turkey
Status: Completed | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Gokhan Gurses, Assistant Professor, Selcuk University
Other Study IDs: SelcukU02
Record Dates: First submitted 2021-06-18; First posted 2021-06-28 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Burnout, Psychological
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to determine the level of burnout in Turkish dentists. The Copenhagen Burnout Inventory of 19 questions will be used to assess burnout; and 4 more about; gender, occupational age, institution and title. All surveys will be conducted online and we plan to reach approximately 400 participants. After the burnout levels are determined, it will be statistically investigated whether there is a difference between the groups according to gender, occupational age, institution and title.

ELIGIBILITY:
Inclusion Criteria:

* Being a dentist who is still working
* Accepted electronically to participate in our study
* Completed and submitted our electronic questionnaires successfully

Exclusion Criteria:

* Did not answer all questions of survey

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Dentist who is still working as a dentist in a health institute.
Sampling Method: Probability Sample
Enrollment: 497 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Participants' burnout levels | 1 month
  Participants' burnout levels will measure by cophenag burnout inventory

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Dentistry Faculty, Selçuklu, Konya, Turkey (Türkiye)